CLINICAL TRIAL: NCT05015686
Title: A Randomized, Blind, Controlled Clinical Trial to Evaluate Safety and Immunogenicity of Live Attenuated Varicella Vaccine After a Two-dose Vaccination Course in Healthy Population Aged ≥13 Years Old
Brief Title: Safety and Immunogenicity of Live Attenuated Varicella Vaccine in Healthy Population Aged ≥13 Years Old
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac (Dalian) Vaccine Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-VZV-4002
Record Dates: First submitted 2021-07-26; First posted 2021-08-20 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Varicella
MeSH Terms: conditions — Chickenpox | interventions — Long-Term Synaptic Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental Group with the immunization course of 0,28 days, 0,42 days or 0,56 days (Experimental): 960 subjects (including 480 children aged 13-17 years and 480 adults aged 18 years and older) will receive two doses of experimental vaccine with the immunization course of 0,28 days, 0,42 days or 0,56 days.
  Interventions: Biological: Live attenuated varicella vaccines manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd
- Control Group (Active Comparator): 960 subjects (including 480 children aged 13-17 years and 480 adults aged 18 years and older) will receive two doses of control vaccine with the immunization course of 0,28 days, 0,42 days or 0,56 days.
  Interventions: Biological: Live attenuated varicella vaccines manufactured by Changchun BCHT Biotechnology Co.,Ltd
- Experimental Group with the immunization course of 0, 70 days (Experimental): 320 subjects (including 160 children aged 13-17 years and 160 adults aged 18 years and older) will receive two doses of the experimental vaccine with the immunization course of 0, 70 days.
  Interventions: Biological: Live attenuated varicella vaccines manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd
- Placebo group (Placebo Comparator): 160 subjects (including 80children aged 13-17 years and 80 adults aged 18 years and older) will receive two doses of the placebo with the immunization course of 0, 70 days.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Live attenuated varicella vaccines manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd — live varicella-zoster virus in 0·5 mL of sucrose, sodium glutamate,sodium chloride,potassium chloride,sodium dihydrogen phosphate, potassium dihydrogen phosphate and injection water per injection
  Arms: Experimental Group with the immunization course of 0,28 days, 0,42 days or 0,56 days
Biological: Live attenuated varicella vaccines manufactured by Changchun BCHT Biotechnology Co.,Ltd — live varicella-zoster virus in trehalose,human serum albumin,sodium glutamate,sucrose,glucose,carbamide,arginine and injection water per injection
  Arms: Control Group
Biological: Live attenuated varicella vaccines manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd — live varicella-zoster virus in 0·5 mL of sucrose, sodium glutamate,sodium chloride,potassium chloride,sodium dihydrogen phosphate, potassium dihydrogen phosphate and injection water per injection
  Arms: Experimental Group with the immunization course of 0, 70 days
Biological: Placebo — Sodium chloride and distilled water
  Arms: Placebo group

SUMMARY:
This a randomized, blind, controlled clinical trial of live attenuated varicella vaccines manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd .The purpose of this study is to evaluate the immunogenicity of a two doses vaccination of investigational vaccine with 0,28 day, 0,42 day and 0,56 day immunization schedule in population aged ≥13 years old.

DETAILED DESCRIPTION:
This study is a randomized, blind, controlled phase # clinical trial in population aged ≥13 years old. The experimental vaccine will be manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd.A total of 2400 subjects aged 13 years and older will be enrolled with1200 subjects in 13 ~ 17 years old group and1200 subjects in 18 years and older group.960 subjects in each age group will be randomly divided into experimental group and control group according to 1:1 ratio,and subjects will receive two doses of vaccine with the immunization course of 0,28 days, 0,42 days or 0,56 days. An additional 240 subjects in each age group will be randomly divided into experimental group and control group according to 2:1 ratio to receive two doses of the experimental vaccine or placebo with the immunization course of 0, 70 days.In addition,400 subjects including 320 people of experimental group in different immunization course according to the difference of age and 80 people of placebo group according to the difference of age will be selected to collect blood about 3ml each time to evaluate immunity persistence of live attenuated varicella vaccines at 3 and 5 years after the whole immunization.

ELIGIBILITY:
Inclusion Criteria:

* Healthy population aged 13 years and above;
* Proven legal identity;
* The subjects and/or guardians can understand and voluntarily sign the informed consent form (For subjects aged 13-17 years, both subjects and guardians need to sign the informed consent form);

Exclusion Criteria:

* History of chickenpox or shingles;
* Axillary temperature >37.0°C;
* Already pregnant (including a positive urine pregnancy test) or are breastfeeding, planning to get pregnant within 6 months;
* History of asthma, history of allergy to the vaccine or vaccine components, or serious adverse reactions to the vaccine, such as urticaria, dyspnea, and angioedema;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc;
* Autoimmune disease or immunodeficiency / immunosuppression;
* Severe chronic diseases, severe cardiovascular diseases,hypertension(adult field measurement: SBP ≥140mmHg or diastolic blood pressure ≥90mmHg)and diabetes that cannot be controlled by drugs, liver or kidney diseases;
* Family history of psychosis,severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Thyroid disease or history of thyroidectomy, asplenia, functional asplenia,asplenia or splenectomy resulting from any condition;
* Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets) or obvious bruising or blood coagulation;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* History of alcohol or drug abuse;
* Receipt of blood products within in the past 3 months;
* Participating in other drug/vaccine clinical trial;
* Receipt of attenuated live vaccines in the past 28 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Onset of various acute or chronic diseases within 7 days prior to the study;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate of the antibody | Day 28 after the whole schedule
  The seroconversion rate of the antibody 28 days among all subjects after the second vaccination.
GMT of the antibody | Day 28 after the whole schedule
  The GMT of the antibody 28 days among all subjects after the second vaccination.

SECONDARY OUTCOMES:
GMI of the antibody | Day 28 after the whole schedule
  GMI of the antibody 28 days among all subjects after the second vaccination.
Seroconversion rate, positive rate, GMT and GMI of the antibody | Day 28,Day 42 and day 56 after the first vaccination
  Seroconversion rate, positive rate, GMT and GMI of the antibody among all subjects on day 28,day 42 and day 56 after the first vaccination.
Incidence of adverse reactions within 0~28 days after each dose | Within 0~28 days after each dose
  Incidence of adverse reactions within 0~28 days after each dose vaccination with immunization course of 0,28 days ,0,42 days and 0,56 days.
Incidence of adverse reactions within 0~14 days after each dose vaccination | Within 0~14 days after each dose
  Incidence of adverse reactions within 0~14 days after each dose vaccination with immunization course of 0,28 days ,0,42 days and 0,56 days
Incidence of grade 3 and above adverse reactions | within 0~28 days after each dose
  Incidence of grade 3 and above adverse reactions within 0~28 days after each dose vaccination with immunization course of 0,28 days ,0,42 days and 0,56 days.
Incidence of serious adverse events | From vaccination to 6 months after the second vaccination
  Incidence of serious adverse events from vaccination to 6 months after the second vaccination with immunization course of 0,28 days ,0,42 days and 0,56 days

CONTACTS AND LOCATIONS:
Overall Officials: Lili Huang, Bachelor, Principal Investigator — Henan Provincial Center for Disease Prevention and Control
Locations (1):
- Yucheng Center for Disease Control and Prevention, Shangqiu, Henan, China